CLINICAL TRIAL: NCT06037317
Title: A Phase Ib, Multi-center, Open-Lable, Dose-Escalation and Dose-Expansion Study of Efficacy and Safety of SY-3505 in Patients With Advanced LTK Fusion-Positive Solid Tumors
Brief Title: A Study of SY-3505 in Patients With Advanced LTK Fusion-Positive Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-3505-I-03
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor
Keywords: SY-3505; Leukocyte receptor tyrosine kinase fusion-positive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation and Dose-expansion (Experimental): In dose-escalation phase, SY-3505 will be given orally in ascending doses (escalation cohort) until the DLT or RP2D is reached.
  In dose-expansion phase, SY-3505 will be given at RP2D in 28-day cycle continuously.
  Interventions: Drug: SY-3505

INTERVENTIONS:
Drug: SY-3505 — LTK tyrosine kinase inhibitor
  Other Names: CT-3505; Ficonalkib

SUMMARY:
This is an open-label, single-arm, multicenter, phase Ib study to evaluate the efficacy and safety of SY-3505 capsule in patients with locally advanced or metastatic, LTK fusion-positive solid tumor who have progressed on or are intolerant to prior standard therapy.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts:

Dose-escalation phase: Participants will be allocated to one of the three dose groups of 500mg, 600mg, or 800mg and receive a single dose of SY-3505 capsules, followed by a 7-day safety observation period and pharmacokinetic (PK) assessment. Subsequently, SY-3505 will be administered once daily in 28-day treatment cycles. This phase is designed to determine the DLTs (Dose-limiting toxicity) and recommended phase II dose (RP2D) and characterize the safety, tolerability and PK of SY-3505 in patients with LTK fusion-positive solid tumors.

Dose-expansion phase: Participants will be assigned to one of the 1-2 dose groups determined during the dose-escalation phase, and receive SY-3505 capsules once daily in 28-day treatment cycles. This phase is designed to evaluate the anti-tumor activity (ORR, DCR and DOR) of SY-3505 in patients with LTK fusion-positive solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for this study:

  1. Age ≥ 18 years at the time of signing the Informed Consent Form (ICF).
  2. Histologically or cytologically confirmed locally advanced (as assessed by the investigator, unresectable tumor or tumor recurrence following standard therapy with evidence of progression [PD] or intolerance to prior therapy) or metastatic solid tumor and failure of standard treatment with evidence of disease progression on imaging.
  3. Agreement to provide a required tumor tissue sample (preferably fresh biopsy tissue or archived tumor tissue within 2 years prior to first dosing) that has been tested by the central laboratory and determined to be positive for LTK gene fusion.
  4. At least one measurable extracranial lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 criteria.
  5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
  6. Expected survival of ≥ 3 months.
  7. Resolution of any treatment-related AEs related to prior anticancer therapy to NCI-CTCAE v 5.0 grade ≤ 1 (excluding toxicities judged by the investigator to be of no safety concern, e.g., hair loss, prior platinum-related grade 2 peripheral neuropathy) before the first dosing.
  8. Organ function levels must meet the following requirements:

     1. No blood products, hematopoietic growth factors (e.g., G-CSF, erythropoietin), or other drugs that correct abnormal blood counts for at least 2 weeks before first dosing and the following blood counts: ANC ≥ 1.5 × 10^9/L, PLT count ≥ 100 × 10^9/L, Hb ≥ 90 g/L.
     2. Liver function: TBIL ≤ 1.5 × upper limit of normal (ULN) in the absence of liver metastases, and AST and ALT ≤ 2.5 × ULN; in the presence of liver metastases, AST and ALT ≤ 5.0 × ULN, and TBIL ≤ 3 × ULN.
     3. Pancreatic function: Serum total amylase ≤ 1.5 × ULN and serum lipase ≤ 1.5 × ULN (subjects with serum total amylase > 1.5 × ULN but with serum lipase within the ULN range may be eligible).
     4. Renal function: Creatinine clearance (Ccr) ≥ 50 mL/min (calculated using the Cockcroft and Gault formula).
     5. Coagulation function: International normalized ratio (INR) and prothrombin time (PT) ≤ 2 × ULN (except for patients receiving anticoagulant therapy).
  9. Able to take oral medications and comply with scheduled visits and related procedures per protocol.
  10. Female subjects of childbearing potential must agree to use highly effective contraception during the entire study period and for at least 3 months after the last dose

Exclusion Criteria:

* Patients who meet any of the following criteria are not eligible for this study:

  1. Carrying known major driver gene mutations other than LTK gene, such as EGFR, MET, ALK, ROS1, NTRK, etc. (Patients with co-mutations may be discussed with the investigator for eligibility).
  2. History of hypersensitivity reactions to any component or excipient of SY-3505 capsules.
  3. Concurrent primary malignancy, with the following exceptions: adequately treated in situ carcinoma, non-melanoma skin cancer, in situ cervical cancer, or in situ breast cancer, and cured malignancies without recurrence for at least 2 years prior to study entry.
  4. Symptomatic primary central nervous system (CNS) tumors, symptomatic CNS metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression. Patients with stable CNS disease (defined as no evidence of progression on imaging for at least 4 weeks prior to first dosing, with all neurological symptoms returned to baseline, and without evidence of new or enlarging brain metastases, and no CNS surgery or radiation treatment within 4 weeks prior to first dosing, and no stereotactic radiosurgery [SRS] within 2 weeks prior to first dosing, and no steroids for at least 2 weeks) are eligible. (Note: Carcinomatous meningitis is not allowed, regardless of clinical stability).
  5. Presence of any of the following conditions or diseases at screening that are inadequately controlled with the best possible medical management:

     1. Active systemic bacterial, viral, or fungal infections.
     2. Pleural effusion, peritoneal effusion, or pericardial effusion that is not controlled after intervention (defined as significant if reaccumulation of fluid requiring drainage occurs within 2 weeks of the prior intervention with associated symptoms).
     3. Poorly controlled diabetes mellitus (defined as fasting blood glucose ≥ 11.1 mmol/L and/or HbA1c ≥ 8%).
     4. Symptomatic hyperthyroidism or hypothyroidism not well controlled by medical management as assessed by the investigator.
     5. Clinically significant electrolyte disturbances (e.g., severe hypocalcemia, hypomagnesemia, hypokalemia) as assessed by the investigator.
     6. Clinically significant gastrointestinal diseases that may interfere with the absorption of study drug (e.g., active ulcerative colitis, Crohn's disease, gastrointestinal ulcers, or major gastrointestinal surgery that might affect drug absorption).
  6. Severe cardiovascular diseases/abnormalities meeting any of the following criteria:

     1. QT interval corrected for heart rate (QTcF) > 470 msec for females or > 450 msec for males as calculated by the Fridericia formula during screening (subjects with suspected drug-induced QTcF prolongation that is assessed by the investigator as safely controllable may be eligible after correction with medication).
     2. Left ventricular ejection fraction (LVEF) < 50%.
     3. Myocardial infarction, unstable angina, or clinically significant arrhythmias (e.g., grade 2 second-degree heart block or third-degree heart block) within 6 months prior to the first dosing.
     4. Class III or IV congestive heart failure as classified by the New York Heart Association (NYHA).
     5. Poorly controlled hypertension, a history of unstable hypertension, or a history of poor compliance with antihypertensive treatment as assessed by the investigator.
  7. Active viral infections or a history of the following:

     1. Active hepatitis B (HBV) infection (defined as HBsAg positive and HBV DNA ≥ 2 × 10^3 IU/mL at screening, unless HBV DNA levels have decreased to < 2 × 10^3 IU/mL after regular antiviral therapy, in which case the patient may be eligible), or active hepatitis C (HCV) infection (HCV RNA > central laboratory ULN) at screening.
     2. HIV positivity at screening or known other immunodeficiency disease.
     3. Previous organ transplantation, hematopoietic stem cell transplantation, or bone marrow transplantation.
  8. Other significant systemic diseases, including but not limited to active pulmonary disease (e.g., active tuberculosis, interstitial lung disease), that, in the investigator's judgment, may affect the interpretation of study results or pose high risks to the patient.
  9. Use of strong CYP3A4 inhibitors or inducers within 2 weeks before the first dosing or during the study period, as follows:

     1. CYP3A4 Inhibitors: Azanavir, Clarithromycin, Erdafitinib, Itraconazole, Ketoconazole, Nafitamone, Letermovir, Saquinavir, Telithromycin, Vinorelbine, Grapefruit (juice).
     2. CYP3A4 Inducers: Carbamazepine, Phenobarbital, Phenytoin, Rifabutin, Rifampicin, St. John's Wort, Rifapentine.
  10. Receipt of any of the following anticancer treatments:

      1. Bone marrow radiation or extensive radiotherapy involving more than 30% of the bone marrow: within 4 weeks before first dosing.
      2. Palliative radiotherapy: within 7 days before first dosing.
      3. Other anticancer treatments such as chemotherapy, targeted therapy (immunotherapy or other antibody therapy), antitumor Chinese medicine, or others: within 2 weeks before first dosing or within 5 half-lives of the treatment (whichever is longer).
  11. Major surgery within 4 weeks before first dosing (major surgery defined as a surgery grade ≥ 3, excluding placement of a central venous catheter, tumor puncture biopsy, and gastrostomy tube placement) or significant traumatic injury that has not fully recovered.
  12. Participation in other clinical studies within 4 weeks before first dosing (except for those that do not use investigational drugs or investigational medical devices; subjects who have discontinued treatment from other clinical studies and are only undergoing follow-up are excluded).
  13. Severe thromboembolic events within 1 year before the first dosing (e.g., cerebrovascular accidents [including transient ischemic attacks], deep vein thrombosis, pulmonary embolism) or a bleeding tendency/risks within 30 days before the first dosing (e.g., significant gastrointestinal bleeding).
  14. Pregnant or lactating women.
  15. Other circumstances, as determined by the investigator, which make the patient unsuitable for participation in this clinical trial, such as other serious acute or chronic diseases that may increase the patient's related risks in the study or laboratory abnormalities that may interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
  Characterization of the safety and tolerability
Incidence of dose limiting toxicities (DLTs) | Escalation Cycle 1 (28 days)
  Maximum Tolerated Dose (MTD) and/or recommended phase 2 dose (RP2D) in Cycle 1

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) for SY-3505 | Protocol-defined time points during Cycle 1 and 2 of treatment (each cycle is 28 days)
  Defined as maximum observed plasma concentration
Pharmacokinetics (Tmax) for SY-3505 | Protocol-defined time points during Cycle 1 and 2 of treatment (each cycle is 28 days)
  Defined as time to maximum plasma concentration
Pharmacokinetics (AUC0-t) for SY-3505 | Protocol-defined time points during Cycle 1 and 2 of treatment (each cycle is 28 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Pharmacokinetics (t½) for SY-3505 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as the apparent plasma terminal phase disposition half-life
Overall Response Rate (ORR) as assessed by RECIST v1.1 | Up to 2 years
  Preliminary anti-tumor activity of SY-3505 in patients with LTK-fusion advanced solid tumor
Disease control rate (DCR) as assessed by RECIST v1.1 | Up to 2 years
  Preliminary anti-tumor activity of SY-3505 in patients with LTK-fusion advanced solid tumor
Duration of response (DOR) as assessed by RECIST v1.1 | Up to 2 years
  Preliminary anti-tumor activity of SY-3505 in patients with LTK-fusion advanced solid tumor

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China